CLINICAL TRIAL: NCT03149497
Title: Anterior Only Surgery for Management of Traumatic Subaxial Cervical Spine Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: arsany botros saleh (Other)
Responsible Party: Sponsor-Investigator, arsany botros saleh, principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: assiutU100
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Traumatic Cervical Spine Instability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- improved anterior approach only in traumatic cervical spine (Active Comparator)
  Interventions: Procedure: anterior approach only in cervical spine trauma
- failed anterior approach only in traumatic cervical spine (Active Comparator)
  Interventions: Procedure: anterior approach only in cervical spine trauma

INTERVENTIONS:
Procedure: anterior approach only in cervical spine trauma — evaluation of efficacy of single approach

SUMMARY:
Classic management of cervical spine sublaxation and dislocation is combined anterior and posterior approach. Unfortunately there are disadvantages for this approach like: increasing morbidity related to each approach, increasing surgical costs, increasing operative time as well as the risk of blood loss.

Anterior approach has the advantages of supine position, less surgical trauma and direct anterior decompression of neural elements. Disadvantages include less mechanical stability and postoperative dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic cases of adult patients with sub axial cervical spine injury presenting to trauma unit of Assiut university hospital

Exclusion Criteria:

* Patients who need cervical corpectomy.
* Pediatric injuries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Radiological analysis | 6 months
  Fusion state by:
  Presence of crossing bone, mobility on motion films and CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt